CLINICAL TRIAL: NCT06273631
Title: Effect of Changes in Carbohydrate Intake Patterns on Glucose Control in Patients with Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Tao (Other)
Responsible Party: Sponsor-Investigator, Yang Tao, professor, Chief physician, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-481
Record Dates: First submitted 2023-02-23; First posted 2024-02-22 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes; Diet Intervention; Glucose Control
Keywords: dietary fiber; autoimmunity; metabolomics; intestinal microbiota; time in range
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- diverse carbohydrate diet (Experimental): Carbohydrate provides 45~55% of total dietary energy, protein 15~20%, and fat 25 ~35%. Among them, 45~50% of carbohydrate supply sources are refined grains, 45~50% of carbohydrate supply sources are whole grains or beans.
  The total energy is divided into 3 meals per day. The breakfast provides 25~30% of total energy, lunch 30~40%，and dinner 30~35%.
  Interventions: Other: diverse carbohydrate diet
- middle carbohydrate diet (Other): Carbohydrate provides 45~55% of total dietary energy, protein 15~20%, and fat 25~35%. 90~95% of the carbohydrate supply comes from refined grains.
  The total energy is divided into 3 meals per day. The breakfast provides 25~30% of total energy, lunch 30~40%，and dinner 30~35%.
  Interventions: Other: middle carbohydrate diet

INTERVENTIONS:
Other: diverse carbohydrate diet — Carbohydrate provides 45~55% of total dietary energy, protein 15~20%, and fat 25 ~35%. Among them, 45~50% of carbohydrate supply sources are refined grains, 45~50% of carbohydrate supply sources are whole grains or beans.
  The total energy is divided into 3 meals per day. The breakfast provides 25~30% of total energy, lunch 30~40%，and dinner 30~35%.
  Arms: diverse carbohydrate diet
Other: middle carbohydrate diet — Carbohydrate provides 45~55% of total dietary energy, protein 15~20%, and fat 25 ~35%. Among them, 90~95% of carbohydrate supply sources are refined grains.
  The total energy is divided into 3 meals per day. The breakfast provides 25~30% of total energy, lunch 30~40%，and dinner 30~35%.
  Arms: middle carbohydrate diet

SUMMARY:
The blood glucose fluctuates greatly in T1DM patients, especially in the middle and late stages of the disease, and carbohydrate (CHO) is the main determinant of postprandial glucose response (PGR). Based on the previous investigation to understand how nutritional habits affect blood glucose control, we will conduct dietary intervention studies in T1DM patients to explore whether the adjustment of dietary pattern is beneficial to blood glucose control, and further explore the relevant mechanism through the detection of related metabolic indicators.

DETAILED DESCRIPTION:
1. Main Objective: To evaluate the effect of changes of carbohydrate intake on glucose control in patients with type 1 diabetes.

1. Primary endpoint: difference of time in range (TIR) between the 2 groups.
2. Secondary endpoint:

1) difference of coefficient of variation (CV), mean amplitude of glycemic excursions (MAGE) , large amplitude of glycemic excursions (LAGE) between the 2 groups; 2) difference of change in HbA1c，GA，1,5-anhydroglucitol (1,5-AG) from baseline between the 2 groups; 3) difference of change in incidence of hypoglycemic events (%), severe hypoglycemia and nocturnal hypoglycemia events from baseline between the 2 groups; 4) difference of change in insulin dose (IU/kg/day) from baseline between the 2 groups.

2. Secondary objective: To explore the possible mechanism of dietary intervention to improve blood glucose control in patients with type 1 diabetes.

1. Effects of dietary intervention on intestinal microenvironment and microflora of type 1 diabetes patients;
2. Effects of dietary intervention on immune function of type 1 diabetes patients;
3. Effects of dietary intervention on metabolomics of type 1 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

1. Those who agree to participate in the study and sign informed consent;
2. Diagnosis of type 1 diabetes mellitus (ADA2024);
3. Age of 18~70 years;
4. Dependent on exogenous insulin therapy, the treatment plan remains unchanged within 2 months (the type of insulin cannot be changed, and the dose can be adjusted according to plasma glucose);
5. Body mass index (BMI) of 18~25kg/m2;
6. HbA1c ≤11%;

Exclusion Criteria:

1. Honeymooners with type 1 diabetes mellitus;
2. Women who are pregnant or plan to become pregnant;
3. Patients who are vegetarians or are undergoing weight loss;
4. Patients who are users of oral hypoglycemic drugs (alpha-glucosidase inhibitors, DPP-IV inhibitors, etc.);
5. Patients who are users of glucocorticoids within 30 days;
6. History of severe food allergy;
7. Patients with acute complications such as DKA or HHS within six months;
8. Patients with gastroparesis, inflammatory bowel disease and other complications;
9. Patients with large albuminuria(albumin-to-creatinine ratio>34.09mg/mmol) and renal insufficiency(creatinine>200umol/L);
10. Patients with uncontrolled hyperthyroidism and hypothyroidism(Uncontrolled hyperthyroidism is defined as abnormal TSH and T4. Uncontrolled hypothyroidism is defined as TSH > 10mIU/L.);
11. History of heart disease, coronary heart disease and arrhythmia;
12. Serious of liver dysfunction (ALT or AST>3 times the upper limit of normal);
13. History of malignant tumors; History of tumors or surgeries affecting digestion and nutrient absorption; Patients with a history of benign tumors, which is judged by the physician to be not suitable;
14. Patients with uncontrolled other immune system diseases or uncontrolled infections;
15. Alcohol abuse, drug abuse, mental disorders or other conditions unfit to be an observer in drug tests;
16. Patients with any disease likely to interfere with study participation or evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time in range (TIR) | Baseline to 2 weeks
  TIR represents percentage of time of glucose levels spent between 3.9 and 10.0 mmol/L based on CGMS. TIR will be compared between the 2 interventions.

SECONDARY OUTCOMES:
Coefficient of variation of blood glucose（CV） | Baseline to 2 weeks
  Reflect glucose fluctuation
Mean amplitude of glycemic excursions（MAGE） | Baseline to 2 weeks
  Reflect glucose fluctuation
Large amplitude of glycemic excursions (LAGE) | Baseline to 2 weeks
  Reflect glucose fluctuation
Change in HbA1c from baseline | Baseline to 14 weeks
  Reflect 2~3 months of glycemic control
Change in GA（glycosylated albumin）from baseline | Baseline to 2 weeks
  Reflect 2~3 weeks of glycemic control
Change in 1,5-anhydroglucitol (1,5-AG) from baseline | Baseline to 2 weeks and to 14 weeks
  Reflect 1~2 weeks of glycemic control
Time above range(TAR) | Baseline to 2 weeks
  TAR represents percentage of time of glucose levels spent over 10.0 mmol/L based on CGMS. TAR will be compared between the 2 interventions.
Time below range(TBR) | Baseline to 2 weeks
  TBR represents percentage of time of glucose levels spent below 3.9 mmol/L based on CGMS. TBR will be compared between the 2 interventions.
Change in total insulin dose from baseline | Baseline to 2 weeks and to 14 weeks
Change in blood lipids from baseline | Baseline to 2 weeks and to 14 weeks
Change in body weight from baseline | Baseline to 2 weeks and to 14 weeks
Daily mean glucose values | Baseline to 2 weeks
Number of participants with severe hypoglycemia and nocturnal hypoglycemia events | Baseline to 2 weeks and to 14 weeks
  Reflects the safety of clinical trials
Change in Incidence of hypoglycemic events from baseline | Baseline to 2 weeks and to 14 weeks
  Reflects the safety of clinical trials
Change in gut microbiota from baseline | Baseline to 2 weeks and to 14 weeks
Change in metabolomics from baseline | Baseline to 2 weeks and to 14 weeks
Change in autoimmunity from baseline | Baseline to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yang, MD/PhD, Principal Investigator — First Affiliated Hospital, Nanjing Medical University, China
Locations (1):
- First Affiliated Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bell E, Binkowski S, Sanderson E, Keating B, Smith G, Harray AJ, Davis EA. Substantial Intra-Individual Variability in Post-Prandial Time to Peak in Controlled and Free-Living Conditions in Children with Type 1 Diabetes. Nutrients. 2021 Nov 19;13(11):4154. doi: 10.3390/nu13114154. PMID 34836409
- [Background] Clark AL, Yan Z, Chen SX, Shi V, Kulkarni DH, Diwan A, Remedi MS. High-fat diet prevents the development of autoimmune diabetes in NOD mice. Diabetes Obes Metab. 2021 Nov;23(11):2455-2465. doi: 10.1111/dom.14486. Epub 2021 Aug 2. PMID 34212475
- [Background] Lejk A, Chrzanowski J, Cieslak A, Fendler W, Mysliwiec M. Effect of Nutritional Habits on the Glycemic Response to Different Carbohydrate Diet in Children with Type 1 Diabetes Mellitus. Nutrients. 2021 Oct 27;13(11):3815. doi: 10.3390/nu13113815. PMID 34836071
- [Background] Thewjitcharoen Y, Wanothayaroj E, Jaita H, Nakasatien S, Butadej S, Khurana I, Maxwell S, El-Osta A, Chatchomchuan W, Krittiyawong S, Himathongkam T. Prolonged Honeymoon Period in a Thai Patient with Adult-Onset Type 1 Diabetes Mellitus. Case Rep Endocrinol. 2021 Sep 1;2021:3511281. doi: 10.1155/2021/3511281. eCollection 2021. PMID 34513096
- [Background] Seidelmann SB, Claggett B, Cheng S, Henglin M, Shah A, Steffen LM, Folsom AR, Rimm EB, Willett WC, Solomon SD. Dietary carbohydrate intake and mortality: a prospective cohort study and meta-analysis. Lancet Public Health. 2018 Sep;3(9):e419-e428. doi: 10.1016/S2468-2667(18)30135-X. Epub 2018 Aug 17. PMID 30122560
- [Background] Jaacks LM, Crandell J, Mendez MA, Lamichhane AP, Liu W, Ji L, Du S, Rosamond W, Popkin BM, Mayer-Davis EJ. Dietary patterns associated with HbA1c and LDL cholesterol among individuals with type 1 diabetes in China. J Diabetes Complications. 2015 Apr;29(3):343-9. doi: 10.1016/j.jdiacomp.2014.12.014. Epub 2014 Dec 31. PMID 25630525
- [Background] Hollowell JG, Staehling NW, Flanders WD, Hannon WH, Gunter EW, Spencer CA, Braverman LE. Serum TSH, T(4), and thyroid antibodies in the United States population (1988 to 1994): National Health and Nutrition Examination Survey (NHANES III). J Clin Endocrinol Metab. 2002 Feb;87(2):489-99. doi: 10.1210/jcem.87.2.8182. PMID 11836274
- [Background] Zhai X, Zhang L, Chen L, Lian X, Liu C, Shi B, Shi L, Tong N, Wang S, Weng J, Zhao J, Teng X, Yu X, Lai Y, Wang W, Li C, Mao J, Li Y, Fan C, Li L, Shan Z, Teng W. An Age-Specific Serum Thyrotropin Reference Range for the Diagnosis of Thyroid Diseases in Older Adults: A Cross-Sectional Survey in China. Thyroid. 2018 Dec;28(12):1571-1579. doi: 10.1089/thy.2017.0715. Epub 2018 Nov 27. PMID 30351201
- [Background] Barouti AA, Bjorklund A, Catrina SB, Brismar K, Rajamand Ekberg N. Effect of Isocaloric Meals on Postprandial Glycemic and Metabolic Markers in Type 1 Diabetes-A Randomized Crossover Trial. Nutrients. 2023 Jul 10;15(14):3092. doi: 10.3390/nu15143092. PMID 37513510
- [Background] Wong K, Raffray M, Roy-Fleming A, Blunden S, Brazeau AS. Ketogenic Diet as a Normal Way of Eating in Adults With Type 1 and Type 2 Diabetes: A Qualitative Study. Can J Diabetes. 2021 Mar;45(2):137-143.e1. doi: 10.1016/j.jcjd.2020.06.016. Epub 2020 Jun 27. PMID 33039330
- [Background] Buehler LA, Noe D, Knapp S, Isaacs D, Pantalone KM. Ketogenic diets in the management of type 1 diabetes: Safe or safety concern? Cleve Clin J Med. 2021 Oct 1;88(10):547-555. doi: 10.3949/ccjm.88a.20121. PMID 34598919
- [Background] Smart CE, Evans M, O'Connell SM, McElduff P, Lopez PE, Jones TW, Davis EA, King BR. Both dietary protein and fat increase postprandial glucose excursions in children with type 1 diabetes, and the effect is additive. Diabetes Care. 2013 Dec;36(12):3897-902. doi: 10.2337/dc13-1195. Epub 2013 Oct 29. PMID 24170749
- [Background] Leow ZZX, Guelfi KJ, Davis EA, Jones TW, Fournier PA. The glycaemic benefits of a very-low-carbohydrate ketogenic diet in adults with Type 1 diabetes mellitus may be opposed by increased hypoglycaemia risk and dyslipidaemia. Diabet Med. 2018 May 8. doi: 10.1111/dme.13663. Online ahead of print. PMID 29737587
- [Background] Vetrani C, Calabrese I, Cavagnuolo L, Pacella D, Napolano E, Di Rienzo S, Riccardi G, Rivellese AA, Annuzzi G, Bozzetto L. Dietary determinants of postprandial blood glucose control in adults with type 1 diabetes on a hybrid closed-loop system. Diabetologia. 2022 Jan;65(1):79-87. doi: 10.1007/s00125-021-05587-0. Epub 2021 Oct 23. PMID 34689215
- [Background] Berry SE, Valdes AM, Drew DA, Asnicar F, Mazidi M, Wolf J, Capdevila J, Hadjigeorgiou G, Davies R, Al Khatib H, Bonnett C, Ganesh S, Bakker E, Hart D, Mangino M, Merino J, Linenberg I, Wyatt P, Ordovas JM, Gardner CD, Delahanty LM, Chan AT, Segata N, Franks PW, Spector TD. Human postprandial responses to food and potential for precision nutrition. Nat Med. 2020 Jun;26(6):964-973. doi: 10.1038/s41591-020-0934-0. Epub 2020 Jun 11. PMID 32528151
- [Background] Kanikarla-Marie P, Jain SK. Hyperketonemia and ketosis increase the risk of complications in type 1 diabetes. Free Radic Biol Med. 2016 Jun;95:268-77. doi: 10.1016/j.freeradbiomed.2016.03.020. Epub 2016 Mar 29. PMID 27036365
- [Background] Bolla AM, Caretto A, Laurenzi A, Scavini M, Piemonti L. Low-Carb and Ketogenic Diets in Type 1 and Type 2 Diabetes. Nutrients. 2019 Apr 26;11(5):962. doi: 10.3390/nu11050962. PMID 31035514
- [Background] Dabek A, Wojtala M, Pirola L, Balcerczyk A. Modulation of Cellular Biochemistry, Epigenetics and Metabolomics by Ketone Bodies. Implications of the Ketogenic Diet in the Physiology of the Organism and Pathological States. Nutrients. 2020 Mar 17;12(3):788. doi: 10.3390/nu12030788. PMID 32192146
- [Background] Zinn C, Lenferna De La Motte KA, Rush A, Johnson R. Assessing the Nutrient Status of Low Carbohydrate, High-Fat (LCHF) Meal Plans in Children: A Hypothetical Case Study Design. Nutrients. 2022 Apr 12;14(8):1598. doi: 10.3390/nu14081598. PMID 35458160
- [Background] Pasmans K, Meex RCR, van Loon LJC, Blaak EE. Nutritional strategies to attenuate postprandial glycemic response. Obes Rev. 2022 Sep;23(9):e13486. doi: 10.1111/obr.13486. Epub 2022 Jun 10. PMID 35686720
- [Background] Saslow LR, Mason AE, Kim S, Goldman V, Ploutz-Snyder R, Bayandorian H, Daubenmier J, Hecht FM, Moskowitz JT. An Online Intervention Comparing a Very Low-Carbohydrate Ketogenic Diet and Lifestyle Recommendations Versus a Plate Method Diet in Overweight Individuals With Type 2 Diabetes: A Randomized Controlled Trial. J Med Internet Res. 2017 Feb 13;19(2):e36. doi: 10.2196/jmir.5806. PMID 28193599
- [Background] Rydin AA, Spiegel G, Frohnert BI, Kaess A, Oswald L, Owen D, Simmons KM. Medical management of children with type 1 diabetes on low-carbohydrate or ketogenic diets. Pediatr Diabetes. 2021 May;22(3):448-454. doi: 10.1111/pedi.13179. Epub 2021 Feb 16. PMID 33470021
- [Background] Turton JL, Raab R, Rooney KB. Low-carbohydrate diets for type 1 diabetes mellitus: A systematic review. PLoS One. 2018 Mar 29;13(3):e0194987. doi: 10.1371/journal.pone.0194987. eCollection 2018. PMID 29596460